CLINICAL TRIAL: NCT01700543
Title: Sidus(TM) Stem-Free Shoulder - A Multi-center, Prospective, Non-controlled Post Market Clinical Follow-up Study.
Brief Title: Sidus(TM) Post Market Clinical Follow-up (PMCF) Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Collaborators: Zimmer, GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2012-01E; 1201E (Other: Zimmer, Inc (Sponsor))
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non-inflammatory Degenerative Joint Disease (NIDJD); Avascular Necrosis; Osteoarthritis; Inflammatory Joint Disease (IJD); Rheumatoid Arthritis
Keywords: Stemless shoulder implant; Osteoarthritis; Rheumatoid Arthritis; Hemi Shoulder Arthroplasty; Total Shoulder Arthroplasty; Prospective; Multi-center; Europe; Non-Controlled; Good Bone Stock
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental: Sidus Shoulder: Patients indicated for hemi or total shoulder arthroplasty with good bone stock who fulfill all inclusion and none of the exclusion criteria.
  Interventions: Procedure: Shoulder Arthroplasty

INTERVENTIONS:
Procedure: Shoulder Arthroplasty — Implantation of the Sidus Stem-Free Shoulder follows standard shoulder replacement procedures.

SUMMARY:
This post market clinical follow-up study is designed to confirm safety and performance of the Sidus Stem-Free Shoulder when used in hemi or total shoulder arthroplasty.

The safety of the implant will be evaluated by monitoring the frequency and incidence of all kinds of adverse events.

The performance will be determined by analyzing the implant survival, overall pain and functional performances (based on Constant & Murley score and ASES score), subject quality of life (EuroQol EQ5D) and radiographic parameters (e.g. radiolucencies, osteolysis, component migration) of study subjects who received the Sidus Stem-Free Shoulder.

The Sidus Stem-Free Shoulder is not approved for use in the US.

DETAILED DESCRIPTION:
This study is a prospective, noncontrolled, multi-center post market clinical follow-up study involving orthopedic surgeons skilled in hemi and total shoulder arthroplasty procedures.

A total number of 160 subjects will be included in the study.

Ethics Committee (EC) approval for each site has to be obtained prior to conducting this study. Sequentially, all eligible patients will be offered study enrollment at each center to avoid potential selection bias. All potential subjects will be required to participate in an informed consent process and sign the EC approved written Informed Consent prior to study enrollment.

The study is designed to be prospective to ensure that the study population is representative of the type of population that the device is intended to treat. Patients will be selected according to the subject selection criteria described in section 8. All subjects will undergo preoperative, intraoperative and immediate postoperative assessments including physical examinations, radiographic evaluations and collection of quality of life metrics. Follow-up evaluations are to be conducted at 3 and 6 months, 1, 2, 5, 7 and 10 years postoperation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 80 years of age, inclusive.
* The patient is skeletally mature.
* Patient is suffering from severe shoulder pain and disability requiring unilateral or bilateral HSA or TSA based on physical exam and medical history.
* Patient has failed conservative treatment.
* Patient meets at least one of the following indications: Osteoarthritis, Posttraumatic arthrosis, Rheumatoid arthritis without humeral metaphyseal defects, Focal avascular necrosis of the humeral head, Previous surgeries of the shoulder that do no compromise the fixation.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved "Informed Consent".

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patients who have any condition which would in the judgement of the Investigator place the patient at undue risk or interfere with the study. Any patient who is institutionalized, or is an known drug abuser, a known alcoholic or anyone who cannot understand what is required of them.
* Patient is known to be pregnant or breastfeeding.
* Patient meets at least one of the contraindications: Soft or inadequate humeral bone (including osteoporosis and extensive avascular necrosis or rheumatoid arthritis) leading to poor implant fixation, Metaphyseal bony defect (including large cysts), Posttraumatic tuberosity non-union, Signs of infection, Irreparable cuff tear, Revision from a failed stemmed prosthesis, Charcot's shoulder (neuroarthropathy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for hemi or total shoulder arthroplasty with good bone stock who fulfill all inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Functional Performance (Constant & Murley Score) | 5 Years
  The Constant & Murley Score (CMS) is a multi-item functional scale assessing pain, ADL, ROM and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively.

SECONDARY OUTCOMES:
Survival (Kaplan-Meier) | 10 years
  The Kaplan-Meier (KM) method is a non-parametric method used to estimate the survival probability from observed survival times (Kaplan and Meier, 1958).
  The survival probability at time ti, S(ti), is calculated as follow:
  S(ti)=S(ti-1)(1-dini)
  Where,
  S(ti-1) = the probability of being alive at ti-1 ni = the number of patients alive just before ti di = the number of events at ti t0 = 0, S(0) = 1

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (8):
- AKH Linz, Linz, Austria
- France (2):
  - Groupe Chirurgical Thiers, Grenoble
  - Centre Hospitalier Universitaire Toulouse, Toulouse
- Germany (3):
  - Charité, Berlin
  - Orthopaedische Chirurgie Muenchen, Munich
  - Gemeinschaftspraxis am Wall, Rinteln
- Azienda Ospedaliera Universitaria Careggi, Florence, Italy
- New Royal Infirmary of Edinburgh, Edinburgh, United Kingdom